CLINICAL TRIAL: NCT02181972
Title: Efficacy and Safety of Gingko Biloba Film-coated Tablets (2 x 60 mg Daily p.o.) in Improving Cognitive Functions and Neuropsychological Functioning of Middle-aged Cognitively Intact Adults: a Double-blind, Placebo-controlled, Parallel Group, Randomised Trial
Brief Title: Efficacy and Safety of Ginkgo Biloba in Middle-aged Cognitively Intact Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1118.2
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Ginkgo Extract

ARMS (2):
- Gingko biloba (Experimental)
  Interventions: Drug: Gingko biloba
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gingko biloba
  Arms: Gingko biloba
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study was to assess the efficacy and safety of Gingko biloba film-coated tablets in improving cognitive function and neuropsychological functioning of middle-aged cognitively intact adults.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy subjects with no known clinically significant pathology as assessed by the investigator
* Mini-Mental State Examination (MMSE) score ≥ 28
* Age range: 40 to 60, inclusive
* Females must test negative for pregnancy
* Clinical laboratory tests must be within normal limits or, if out of normal range, clinically acceptable to the Investigator
* Urine drug screen for illicit drugs must be negative at screening
* Subjects must have given written informed consent in accordance with ICH-GCP (International Conference on Harmonization - Good Clinical Practice) and local laws and regulations

Exclusion Criteria:

* Any serious disorder that may interfere with his/her participation in the trial and the evaluation of the safety of the test drug
* Pre-treatment and/or concomitant treatment with any drug that may influence the trial symptomatology and may interfere with the evaluation of cognitive function
* Alcohol and drug abuse according to DSM-IV (Diagnostic and Statistics Manual, Version IV)
* Individuals drinking more than 6 cups of coffee or tea/day
* Individuals smoking more than 10 cigarettes/day
* Subjects who in the opinion of the investigator are heavy users of other tobacco or nicotine products
* Subjects currently taking a cognition enhancing substance, including any Ginkgo or ginseng product
* Any subject regularly taking a medication who might stop doing so at some time during the active dosing phase, if the medication is deemed by the investigator to influence the outcome of the trial
* Female subjects of child-bearing age who are not using adequate means of birth control
* Pregnancy and/or lactation
* Any subject who, according to the Investigator, is unable to perform the CDR cognitive tests or the neuropsychological tests in a satisfactory and consistent manner
* Relevant allergy or known hypersensitivity to the investigational product or its excipients
* Individuals under anticoagulant treatment
* Individuals with a current disorder likely to modify computerised cognitive testing
* Individuals having a history of cancer (any type, excluding surgically removed and treated basal cell carcinoma)
* Clinically significant and not treated thyroid disease
* Participation in another clinical trial within the last 3 months prior to the start of the study and concurrent participation in another clinical trial

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2002-05; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of the cognitive test/CDR (Cognitive Drug Research) factor "Power of Attention) | pre-dose and 2, 4, 6 hours post-dosing at baseline and day 56

SECONDARY OUTCOMES:
Changes from baseline in CDR factors | pre-dose and 2, 4, 6 hours post-dosing at baseline, days 28 and 56
Changes from baseline in Stroop Colour and Word Test | Baseline and day 56
Changes from baseline in the Selective Reminding Test | Baseline and day 56
Changes from baseline in the Trail Making Test (Part A and B) | Baseline and day 56
Number of patients with adverse events | up to 56 days
Number of patients with clinically significant changes in vital signs | Baseline, days 28 and 56
Number of patients with abnormal changes in laboratory parameters | Baseline and day 56
Assessment of tolerability by subject on a 4-point scale | Days 28 and 58
Assessment of tolerability by investigator on a 4-point scale | Days 28 and 58